CLINICAL TRIAL: NCT06418360
Title: Evaluation of The Efficacy of TECAR Therapy in Patients With Knee Osteoarthritis
Brief Title: Efficacy of TECAR Therapy in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-23-3792
Record Dates: First submitted 2024-05-06; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis; Energy Transfer Capacitative and Resistive Therapy
Keywords: knee pain, osteoarthritis, capacitative and resistive energy transfer therap
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical therapy (CPT) (Experimental): Group 1 (HP, TENS, knee isometric and theraband exercise) to painful side knee area, two weeks, five times a week, 10 sessions.
  Interventions: Device: conventional physical therapy; Transcutaneous Electrical Nerve Stimulation, hotpack
- conventional physical therapy (CPT) and TECAR therapy (Experimental): Group 2 (HP, TENS, knee isometric and theraband exercise) 10 sessions, two weeks, five times a week and in addition TECAR therapy, to painful side knee quadriceps and peripatellar area, three times a week for two weeks, for a total of 6 sessions.
  Interventions: Device: TECAR

INTERVENTIONS:
Device: TECAR — Transfer Energy Capacitative and Resistive Therapy
  Arms: conventional physical therapy (CPT) and TECAR therapy
Device: conventional physical therapy; Transcutaneous Electrical Nerve Stimulation, hotpack — 10 sessions of HP and TENS for two weeks, five times a week. HP was applied to the painful knee area for 20 minutes using a heating pad for superficial heating purposes. TENS was applied to the painful knee area for 20 minutes at 80 Hz frequency
  Arms: conventional physical therapy (CPT)

SUMMARY:
Objective: The aim of the present study was to investigate the treatment efficacy of TECAR therapy, a modern application that has been increasingly used in recent years, compared to conventional physical therapy applications in the treatment of knee osteoarthritis, according to the evaluation of the clinical findings of patients.

Methods: A total of 54 patients, aged between 40 and 75 years, were randomly divided into two groups. Both groups received CPT. Group 2 received TECAR therapy in addition to CPT, applied three times a week for two weeks, for a total of 6 sessions. All patient's knee joint range of motion (ROM) was measured goniometrically, isometric quadriceps muscle strength was measured, and pain levels were assessed using the Visual Analog Scale (VAS), and disability levels were assessed using the Western Ontario and McMaster Universities Arthritis Index (WOMAC) before treatment, at the end of treatment, at 1 month, and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* 3 months of conservative treatment for unresponsive knee pain
* Kellgren-Lawrence grade 2-3 on radiographic evaluation
* Agreed to participate in the study.

Exclusion Criteria:

* History of physical therapy (electrotherapy/exercise) in the past 3 months
* Intra-articular injection therapy in the past 3 months,
* History of surgery or trauma to the affected knee
* Inflammatory or neurological disease affecting the lower extremities
* Active vasculitis or severe peripheral vascular disease
* Pregnancy or lactation
* Diagnosed restless legs syndrome
* Neoplasia
* Local sensory impairment,
* Local or systemic acute infections
* Severe osteoporosis
* Pacemaker
* Psychiatric disorder and cognitive impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Before and the after treatment 0th day , 1th month, 3rd month
  0 min , 10 is maximum pain score
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Before and the after treatment 0th day, 1th month, 3rd month
  This 24-item index comprises three subscales: pain, stiffness, and physical function, each measured on a five-point Likert scale ranging from "none" to "extreme."
Range of Motion (ROM) | Before and the after treatment 0th day, 1th month, 3rd month
  Flexion and extension of the knee joint were measured using a universal goniometer relative to reference points.

SECONDARY OUTCOMES:
The Diers Myoline Isometric Muscle Strength Measurement System | Before and the end of treatment 0th day, 1th month, 3rd month
  quadriceps muscle Isometric Strength Measure: Increased isometric muscle strength is an indicator of recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Özge TEZEN, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
participant data will not share